CLINICAL TRIAL: NCT03479892
Title: A Randomised, Double-blinded, Multiple-dose, Dose-escalation Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC0194-0499 in Subjects With Overweight or Obesity
Brief Title: A Research Study Looking at a New Study Medicine (NNC0194-0499) for Weight Control in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9499-4287; U1111-1193-7228 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-03-09; First posted 2018-03-27 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0194-0499 (Experimental): Participants will receive increasing doses of NNC0194-0499. The treatment period from first treatment (Day 1) to end of the treatment (Day 85) will be 12 weeks.
  Interventions: Drug: NNC0194-0499
- Placebo (Placebo Comparator): Participants will receive NNC0194-0499 matched placebo. The treatment period from first treatment (Day 1) to end of the treatment (Day 85) will be 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC0194-0499 — Participants will receive NNC0194-0499 (s.c., in a lifted fold of the abdominal skin) injection once weekly at increasing doses of 3.0 mg, 9.0 mg, 27 mg, 60 mg, or 120 mg. Each participant will only be given one dose level.
  Dose escalation will proceed to the next planned dose level if there are no safety concerns raised by the investigator or by the trial safety group.
  Arms: NNC0194-0499
Drug: Placebo — Participants will receive once weekly injections of NNC0194-0499 matched placebo.
  Arms: Placebo

SUMMARY:
This study looks at a new study medicine for weight control in people with overweight or obesity. The aim of this study is to see if the study medicine is safe for people to take. The study also looks at how fast the body removes the study medicine. The participants will either get NNC0194-0499 (the study medicine) or placebo (a formula that looks like the medicine but does not have active ingredients). Which treatment the participants get is decided by chance. The participants will get 1 or more injections into the skin of stomach area once each week for 12 weeks. The study will last for about 4 to 5 months. The participants will have 18 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male aged 22-55 years (both inclusive) or female aged 22-45 years (both inclusive) at the time of signing informed consent
* Female must have regular menstrual cycle(defined as 24-35 days between 1st day of menses for two most recent menstrual periods, self-reported)
* Female must have bilateral tubal ligation or must be willing to use non-hormonal intrauterine device or diaphragm /cervical cap with spermicide in combination with condom for male partner(s)
* Body mass index (BMI) between 27.0 and 39.9 kg/sqm (both inclusive). Overweight should be due to excess adipose tissue, as judged by the investigator
* Considered by the investigator to be generally healthy based on the medical history, physical examination, and the results of vital signs, ECG, and clinical laboratory tests performed during the screening visit

Exclusion Criteria:

* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol
* Use of prescription or non-prescription medicinal products including herbal products and non-routine vitamins, within 2 weeks prior to screening. Mild painkillers are allowed until 24 hours prior to screening
* History or presence of bone disease or otherwise increased risk of bone fracture as evaluated by dual-energy x-ray absorptiometry and as judged by the investigator

Ages: 22 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | From first administration of NNC0194-0499 (Day 1) to follow-up (Day 112)
  count of events

SECONDARY OUTCOMES:
Change in heart rate | Baseline (Day 1), Follow-up (Day 112)
  measured in beats per minute
Change in biochemistry | Baseline (Day -1), Follow-up (Day 112)
  Parameters: Calcium (total), Chloride, Magnesium, Phosphate (inorganic), Potassium, Sodium, Urea (blood urea nitrogen, BUN), Uric acid, Alanine aminotransferase (ALT), Alkaline phosphatase (ALP), Amylase, Aspartate aminotransferase (AST), Creatinine kinase (CK, total), Gamma glutamyltransferase (GGT), Lactase dehydrogenase, Lipase, Albumin, Bicarbonate, Bilirubin (total), Creatinine, High sensitivity C-reactive protein (hsCRP) and Total protein in SI units
Change in haematology | Baseline (Day -1), Follow-up (Day 112)
  Parameters: Erythrocytes, Reticulocytes, Thrombocytes, Leucocytes (total), Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils, Haemoglobin, Haematocrit, Mean corpuscular volume (MCV) and Mean corpuscular haemoglobin concentration (MCHC) in SI units
Change in fibrinogen | Baseline (Day -1), Follow-up (Day 112)
  measured in g/L
Change in prothrombin time read as international normalised ratio (INR) | Baseline (Day -1), Follow-up (Day 112)
Change in activated partial thromboplastin time (APTT) | Baseline (Day -1), Follow-up (Day 112)
  measured in seconds
Changes in electrocardiogram (ECG) | Baseline (Day 1), Follow-up (Day 112)
  Parameters: RR interval, PR interval, QRS interval, QT interval and QTcF interval in SI units
Number of injection site reactions | From baseline (Day 1) to follow-up (Day 112)
  count of injection site reactions
Occurrence of anti-NNC0194-0499 antibodies | From baseline (Day 1) to follow-up (Day 112)
t½,SS: the terminal serum half-life of NNC0194-0499 at steady state | From last dose (Day 78, pre-dose) until the follow-up (Day 112)
  Calculated based on serum concentrations of NNC0194-0499
Cmax,SS: the maximum concentration of NNC0194-0499 in serum at steady state | From last dose (Day 78, pre-dose) until the follow-up (Day 112)
  Calculated based on serum concentrations of NNC0194-0499
tmax,SS: the time to maximum concentration of NNC0194-0499 in serum at steady state | From last dose (Day 78, pre-dose) until the follow-up (Day 112)
  Calculated based on serum concentrations of NNC0194-0499
CL/F SS: the apparent total serum clearance of NNC0194-0499 at steady state | From last dose (Day 78, pre-dose) until the follow-up (Day 112)
  Calculated based on serum concentrations of NNC0194-0499
Change in systolic blood pressure | Baseline (Day 1), Follow-up (Day 112)
  measured in mmHg
Change in diastolic blood pressure | Baseline (Day 1), Follow-up (Day 112)
  measured in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://www.novonordisk-trials.com